CLINICAL TRIAL: NCT06428786
Title: The Effect of Polycystic Ovary Syndrome Phenotypes on Quality of Life and Sexual Function
Acronym: PCOS
Status: Completed | Type: Observational
Sponsor: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mujde Can Ibanoglu, Assoc. Prof, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Other Study IDs: 02/08 28.02.2024
Record Dates: First submitted 2024-05-18; First posted 2024-05-24 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Polycystic Ovary; Depression; Sexual Dysfunction
Keywords: Female Sexual Function Index; phenotypes; polycystic ovary syndrome; The Beck Depression Inventory; Quality of life
MeSH Terms: conditions — Polycystic Ovary Syndrome; Depression; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Phenotype A: PHENOTYPE A: Hyperandrogenism + Ovulatory Dysfunction + Polycystic ovary morphology 44 participants
  Interventions: Other: Female Sexual Function Index
- Phenotype B: PHENOTYPE B: Hyperandrogenism + Ovulatory Dysfunction 44 participants
  Interventions: Other: Female Sexual Function Index
- Phenotype C: PHENOTYPE C: Hyperandrogenism + Polycystic ovary morphology 44 participants
  Interventions: Other: Female Sexual Function Index
- Phenotype D: PHENOTYPE D: Ovulatory Dysfunction + Polycystic ovary morphology 44 participants
  Interventions: Other: Female Sexual Function Index

INTERVENTIONS:
Other: Female Sexual Function Index — As part of the study, data on the socio-demographic characteristics of the individuals is collected by means of personal interviews using a questionnaire. The results of laboratory tests required for the diagnosis of PCOS will be taken from hospital records. The Female Sexual Function Index (FSFI), the Beck Depression Inventory and the KF-36 quality of life assessment form will be completed in person and the total scores will be analyzed taking into account four different PCOS phenotypes.
  Other Names: Beck Depression Inventory; Short Form 36

SUMMARY:
This study was planned to examine whether different phenotypes of PCOS have an effect on quality of life, depression inventory and sexual function.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrinologic pathology in women of reproductive age. Although the prevalence varies according to race, ethnicity and geographical region, it averages between 5-10%. The so-called Rotterdam criteria are: 1. Oligo- and/or anovulation, 2. Clinical and/or biochemical signs of hyperandrogenism, 3. Polycystic ovarian morphology on ultrasound, 4. Other conditions causing or associated with androgen elevation must be ruled out before a diagnosis of PCOS is made. Treatment needs, types and options vary according to phenotypic characteristics. The OD+HA+PKOM phenotype is considered a complete (classic) phenotype according to the Rotterdam classification and has the highest rate. Other phenotypes according to the Rotterdam criteria can be OD+HA (non-PCO phenotype), HA+PKOM (ovulation phenotype) or OD+PKOM (non-HA phenotype). Clinical pictures (phenotype A: HA + OD + PCOM; phenotype B: HA + OD; phenotype C: HA + PCOM and phenotype D: OD + PCOM). According to the Rotterdam criteria, endocrine and metabolic abnormalities are lowest in the OD+PCOM group among these 4 different phenotypes. The prevalence and distribution characteristics of metabolic abnormalities (insulin resistance, metabolic disease pattern and glucose intolerance) did not differ significantly between the 4 groups. Therefore, metabolic abnormalities and distribution characteristics are not used to differentiate the different clinical PCOS phenotypes.

Studies have shown that the "classic" PCOS group (phenotypes A and B) is more strongly associated with marked menstrual irregularity, elevated insulin levels and risk of metabolic syndrome; body mass index and obesity compared to the non-classic or non-hyperandrogenic PCOS phenotypes (phenotypes C and D).

There are numerous studies on whether phenotypic differences are based on ethnicity. Studies have shown that African-American women and women of Hispanic origin are more prone to obesity and the development of metabolic syndrome, while Middle Eastern women and women of Mediterranean origin are more prone to hirsutism. PCOS symptoms such as clinical hyperandrogenism, anovulation and menstrual irregularities can lead to a reduced quality of life, depression, mood disorders and sexual dysfunction. The physical, emotional and environmental scores were significantly lower in Group A patients compared to the other PCOS groups and the control group. The Short Form 36 (SF 36), which has the characteristics of a general scale among quality of life scales and provides broad measurement, was developed and put into use by the Rand Corporation in 1992. The scale was designed to be short and easy to administer and has a wide range of applications. The main feature of the SF-36, whose psychometric properties and scope have been expanded, is that it is a self-report scale that includes items on physical functioning, social functioning, role limitations related to physical functioning, role limitations related to emotional problems, mental health, energy/vitality, pain, and general perception of health.

The relationship between the severity of depressive symptoms and the different PCOS phenotypes is controversial. The Beck Depression Inventory (BDI-II), developed by Dr. Aaron T. Beck, is a questionnaire with 21 multiple-choice questions that can be used to measure the severity of depression. Scores ≥17 indicate severe depression requiring treatment.The depression inventory scores were higher in PCOS patients with infertility problems. A study found that there was no difference in depression scores between infertile and fertile groups.

The Female Sexual Function Index (FSFI) inventory was used to assess sexual dysfunction in obese PCOS patients. The Female Sexual Function Index was developed in 2000 to assess sexual function in women. The scale consists of 19 items and has 6 sub-dimensions: Pleasure, Arousal, Lubrication, Orgasm, Satisfaction and Pain. The scale reflects women's sexual functioning in the past month by calculating 6 subgroup scores and the FSFI score. The FSFI score is calculated by adding the subgroup scores. The Female Sexual Function Index has proven to be a valid and reliable tool for measuring sexual function in Turkish women.

Based on this information, the aim of this study was to investigate whether different phenotypes of PCOS have an impact on quality of life, depression inventory and sexual function.

ELIGIBILITY:
Inclusion Criteria:

* least 1 year after menarche
* over 18 years old
* Patients who have given verbal and written informed consent will be included.

Exclusion Criteria:

* under 18 years of age
* Endocrine disorders such as hyperprolactinemia, Cushing's syndrome, congenital adrenal hyperplasia, thyroid disorders
* Neuromuscular, hepatic, pancreatic or gastrointestinal diseases
* Users of hormone preparations such as antiandrogens, antidiabetics, glucocorticoids, insulin sensitizers, lipid regulators

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sexually active people who are cared for at the PCOS Clinic of Etlik Zübeyde Hanım Gynecology Training and Research Hospital form the study group.
  The study involves 176 subjects who agreed to participate in the study and accepted the informed consent verbally and in writing.
  The ESHRE/ASRM 2023 guidelines will be used as a basis and those who fulfill both criteria below will be included in the PCOS group:
  1. Oligo and/or anovulation*
  2. Clinical and/or biochemical hyperandrogenism
  3. Polycystic ovarian morphology or AMH elevation
  Definition of the phenotype groups: PCOS has been categorized into 4 phenotypes:
  Phenotype A: Hyperandrogenism + ovarian dysfunction + PCOM PHENOTYPE B: HA+OD PHENOTYPE C: HA+PCOM PHENOTYPE D: OD+PKOM were grouped as.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Effect of PCOS phenotypes on SF-36. | 6 months
  The aim of this study was to investigate whether different phenotypes of PCOS have an impact on quality of life, depression inventory and sexual function.
Effect of PCOS phenotypes on FSFI. | 6 months
  The aim of this study was to investigate whether different phenotypes of PCOS have an impact on quality of life, depression inventory and sexual function.
Effect of PCOS phenotypes on Beck Deppression scale | 6 months
  The aim of this study was to investigate whether different phenotypes of PCOS have an impact on quality of life, depression inventory and sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Mujde Can Ibanoglu, Principal Investigator — Ankara Etlik Zubeyde Hanım Women's Health Training and Research Hospital, Ankara, Turkey.
Locations (1):
- Etlik Zübeyde Hanım, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tian X, Ruan X, Du J, Cheng J, Ju R, Mueck AO. Sexual function in Chinese women with different clinical phenotypes of polycystic ovary syndrome. Gynecol Endocrinol. 2023 Dec;39(1):2221736. doi: 10.1080/09513590.2023.2221736. PMID 37302412
- [Result] Yilmaz M, Isaoglu U, Delibas IB, Kadanali S. Anthropometric, clinical and laboratory comparison of four phenotypes of polycystic ovary syndrome based on Rotterdam criteria. J Obstet Gynaecol Res. 2011 Aug;37(8):1020-6. doi: 10.1111/j.1447-0756.2010.01478.x. Epub 2011 Apr 12. PMID 21481088